CLINICAL TRIAL: NCT01359566
Title: A Randomized, Double Blind, Placebo-Controlled Efficacy and Safety Study of Arbaclofen Placarbil in Subjects With Spasticity Due to Multiple Sclerosis
Brief Title: Efficacy and Safety of Arbaclofen Placarbil in Subjects With Spasticity Due to Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XP-B-089; NCT01360489 (obsolete NCT alias)
Record Dates: First submitted 2011-05-22; First posted 2011-05-24 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — arbaclofen placarbil; BID protein, human; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arbaclofen placarbil 15 mg BID (Active Comparator): Arbaclofen placarbil (XP19986 SR4) 15 mg every morning and every evening
  Interventions: Drug: Arbaclofen placarbil 15 mg BID
- Arbaclofen placarbil 30 mg BID (Active Comparator): Arbaclofen placarbil (XP19986 SR4) 30 mg every morning and every evening
  Interventions: Drug: Arbaclofen placarbil 30 mg BID
- Arbaclofen placarbil 45 mg BID (Active Comparator): Arbaclofen placarbil (XP19986 SR4) 45 mg every morning and every evening
  Interventions: Drug: Arbaclofen placarbil 45 mg BID
- Placebo (Placebo Comparator): Placebo every morning and every evening
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arbaclofen placarbil 15 mg BID — arbaclofen placarbil 15 mg BID
  Other Names: XP19986 SR4
  Arms: Arbaclofen placarbil 15 mg BID
Drug: Placebo — Placebo for arbaclofen placarbil 15, 30 and 45 mg BID
  Other Names: Sugar Pill
  Arms: Placebo
Drug: Arbaclofen placarbil 30 mg BID — arbaclofen placarbil 30 mg BID
  Other Names: XP19986 SR4
  Arms: Arbaclofen placarbil 30 mg BID
Drug: Arbaclofen placarbil 45 mg BID — arbaclofen placarbil 45 mg BID
  Other Names: XP19986 SR4
  Arms: Arbaclofen placarbil 45 mg BID

SUMMARY:
To evaluate the efficacy of three doses of XP19986 (arbaclofen placarbil) compared to placebo for the treatment of spasticity in subjects with multiple sclerosis (MS).

ELIGIBILITY:
Inclusion Criteria:

1. Has multiple sclerosis (MS) based on Poser or McDonald Criteria (all subtypes of MS will be accepted, including relapsing remitting, primary or secondary progressive, if disease is stable per exclusion criteria).
2. Maximum Ashworth Score Scale score of ≥ 2 in at least one of the following muscle groups on either side of the body: hip abductors/adductors, knee flexors/extensors, ankle flexors/extensors.
3. Expanded Disability Status Scale (EDSS) rating between 3.0-8.0 inclusive.
4. If a subject is on disease modifying MS treatment, the dosage, frequency, and route of administration must be stable for at least 30 days before screening and is expected to be stable throughout the study.
5. Spasticity Disability Rating of 2 or higher at Baseline.
6. Willing to discontinue and refrain from using for the duration of the study drugs for the treatment of spasticity or likely to affect spasticity (including, but not limited to, baclofen, tizanidine, diazepam, clonazepam, metaxalone, dantrolene, cyclobenzaprine, carisoprodol, clonidine, vigabatrin, valproic acid and cannabis).

Exclusion Criteria:

1. Spasticity due to neurological disorder other than MS or other conditions that may confound the assessment of spasticity.
2. Subject has clinically evident muscle contractures resulting in irreversible spasticity in lower extremities.
3. Subjects who have suffered an acute relapse of MS (as determined by the Investigator) within 90 days prior to Screening, or have had more than 1 relapse within the year prior to Screening
4. Botulinum toxin injection within 6 months of Screening or has current residual associated side effects at Screening.
5. Subjects receiving concomitant medication from more than one of the following three drug classes: (Antiepileptic drugs, Tricyclic anti-depressants and Opioids)
6. Subjects on the following medications, at doses above the specified limits, are excluded if they cannot maintain a level within these limits

   * Gabapentin ≤ 1800 mg per day or pregabalin ≤ 150 mg per day
   * Amitriptyline ≤ 75 mg per day or nortriptyline ≤ 75 mg per day
   * Opioids ≤ 30 mg morphine equivalents per day.
7. Evidence of unstable or severe systemic illness, including but not limited to: Cardiovascular disease (e.g., chronic ventricular arrhythmia, unstable angina or CHF), respiratory disease (e.g., sleep apnea, COPD requiring oxygen therapy or hospitalization in last year), endocrine disease, hepatic disease (e.g., chronic active hepatitis), renal disease, or immunodeficiency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2011-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Maximum Ashworth Scale score (6 hour post-dose time point) | 10-weeks
  numerical score
Patient Global Impression of Change (PGIC) score | 10-weeks
  numerical score

SECONDARY OUTCOMES:
Change in the overall Modified PRISM score | Weeks 4, 6, 10
  Variables
Change in weekly average severity of pain score associated with muscle spasm. | Week 10
  numerical score
Change in weekly average VAS score of sleep quality | Week 10
  numerical score

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Indivior Inc.
Locations (28):
- United States (28):
  - XenoPort Clinical Site, Phoenix, Arizona
  - XenoPort Clinical Site, Tucson, Arizona
  - XenoPort Clinical Site, Berkeley, California
  - XenoPort Clinical Site, San Diego, California
  - XenoPort Clinical Site, Denver, Colorado
  - XenoPort Clinical Site, Port Charlotte, Florida
  - XenoPort Clinical Site, Sarasota, Florida
  - XenoPort Clinical Site, St. Petersburg, Florida
  - XenoPort Clinical Site, Tampa, Florida
  - XenoPort Clinical Site, Lake Barrington, Illinois
  - XenoPort Clinical Site, Indianapolis, Indiana
  - XenoPort Clinical Site, Lenexa, Kansas
  - XenoPort Clinical Site, Lexington, Kentucky
  - XenoPort Clinical Site, Bingham Farms, Michigan
  - XenoPort Clinical Site, Detroit, Michigan
  - XenoPort Clinical Site, Toms River, New Jersey
  - XenoPort Clinical Site, Albuquerque, New Mexico
  - XenoPort Clinical Site, Albany, New York
  - XenoPort Clinical Site, Patchogue, New York
  - XenoPort Clinical Site, Plainview, New York
  - XenoPort Clinical Site, Asheville, North Carolina
  - XenoPort Clinical Site, Akron, Ohio
  - XenoPort Clinical Site, Franklin, Tennessee
  - XenoPort Clinical Site, Nashville, Tennessee
  - XenoPort Clinical Site, San Antonio, Texas
  - XenoPort Clinical Site, Vienna, Virginia
  - XenoPort Clinical Site, Seattle, Washington
  - XenoPort Clinical Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Command Clinical Research Trial Website — https://www.ispot.tv/ad/7LIc/command-clinical-research-study-ms-spasticity